CLINICAL TRIAL: NCT02250573
Title: An Open-study to Investigate the Safety and Efficacy of Replenine®-VF in Haemophilia B Subjects Undergoing Surgery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: R9VFSUR
Record Dates: First submitted 2014-09-02; First posted 2014-09-26 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Haemophilia B
MeSH Terms: conditions — Hemophilia B

ARMS (1):
- Replenine®-VF (Experimental)
  Interventions: Biological: Replenine®-VF (High Purity Factor IX)

INTERVENTIONS:
Biological: Replenine®-VF (High Purity Factor IX)

SUMMARY:
The main objectives of this study were to investigate the safety and efficacy of Replenine®-VF administered in appropriate dosage by bolus infusion to prevent bleeding and achieve haemostasis in subjects with haemophilia B undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe haemophilia B undergoing major surgery requiring an in-patient stay of generally 5 to 10 days.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-12; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Incremental recovery for Factor IX | 90 min post-dose
  Incremental recovery is defined as peak rise in plasma Factor IX levels divided by Factor IX dose in IU/KG

CONTACTS AND LOCATIONS:
Locations (5):
- Samodzielny Publiczny Zaklad Opieki Zdrowotnej nad Matka I Dzieckiem, ul. Krysiewicza 7/8., Poznan, Poland
- Romania (2):
  - Institutul National de Haemtologie, 2-8 Constantin Caracas Str., Bucharest
  - Spitalul de urgenta pentru copii "Louis Turcana", Str. losef Nemoianu 2., Timișoara
- Russia (2):
  - Kirov Research Institute of Haematology, 72 Krasnoarmeyskaya ul., Kirov
  - Haematology Centre, Russian Academy if Medical Sciences, 4a Novozykovsky Proezed., Moscow

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk